CLINICAL TRIAL: NCT06630832
Title: Impact of Partial and Full Cooling Applied During Prescribed Rest Breaks to Mitigate Increases in Physiological Strain During Prolonged Work in Hot Environments.
Brief Title: Initial Stay Times and Heat Mitigation Controls for Uncompensable Occupational Heat Stress - Part III
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Ottawa (Other)
Responsible Party: Principal Investigator, Glen P. Kenny, Full Professor, University of Ottawa
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: HEPRU-2024-09-B
Record Dates: First submitted 2024-10-04; First posted 2024-10-08 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-06

CONDITIONS: Body Temperature Changes; Heat Stress; Heat Exposure; Heat Fatigue; Work Related Stress; Hyperthermia
Keywords: Heat strain; Thermoregulation; Exercise; Core temperature; Occupational heat stress; Uncompensable heat stress; Aging
MeSH Terms: conditions — Body Temperature Changes; Heat Stress Disorders; Occupational Stress; Hyperthermia; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- No cooling (Active Comparator): Participants perform a continuous moderate-intensity work bout (metabolic rate of ~200 W/m2) until core temperature reaches 38.0°C (equivalent to a 1°C increase in body core temperature above resting levels), which is immediately followed by intermittent work using a 1:3 work-rest allocation, starting with a 45 min rest break followed by a 15 min work bout for an additional 180-min of work without cooling.
  Interventions: Other: Simulated work in the heat with no cooling during rest breaks
- Partial cooling (Experimental): Participants perform a continuous heavy-intensity work bout (metabolic rate of ~200 W/m2) until core temperature reaches 38.0°C (equivalent to a 1°C increase in body core temperature above resting levels), which is immediately followed by intermittent work using a 1:3 work-rest allocation, starting with a 45 min rest break followed by a 15 min work bout for an additional 180-min of work with partial cooling equivalent to sitting in a shaded space (WBGT 24°C; 31.7°C and 35% RH) such as under a tree with a light breeze (simulated with pedestal fan fixed at ~2 m/s).
  Interventions: Other: Simulated work in the heat with partial cooling during rest breaks
- Full cooling (Experimental): Participants perform a continuous heavy-intensity work bout (metabolic rate of ~200 W/m2) until core temperature reaches 38.0°C (equivalent to a 1°C increase in body core temperature above resting levels), which is immediately followed by intermittent work using a 1:3 work-rest allocation, starting with a 45 min rest break followed by a 15 min work bout for an additional 180-min of work with full cooling equivalent to sitting in air-conditioned space (e.g., room or vehicle) maintained at 22°C and 35% RH (equivalent WBGT of 16°C).
  Interventions: Other: Simulated work in the heat with full cooling during rest breaks

INTERVENTIONS:
Other: Simulated work in the heat with no cooling during rest breaks — Young and older adults will not undergo cooling during rest breaks applied during the implementation of work-rest allocations over the duration of a 180-min work period following a continuous work bout to 38.0°C (equivalent to a 1°C increase in body core temperature above resting levels).
  Arms: No cooling
Other: Simulated work in the heat with partial cooling during rest breaks — Young and older adults will not undergo partial cooling during rest breaks applied during the implementation of work-rest allocations over the duration of a 180-min work period following a continuous work bout to 38.0°C (equivalent to a 1°C increase in body core temperature above resting levels).
  Arms: Partial cooling
Other: Simulated work in the heat with full cooling during rest breaks — Young and older adults will not undergo full cooling during rest breaks applied during the implementation of work-rest allocations over the duration of a 180-min work period following a continuous work bout to 38.0°C (equivalent to a 1°C increase in body core temperature above resting levels).
  Arms: Full cooling

SUMMARY:
Occupational heat stress directly threatens workers' ability to live healthy and productive lives. Heat exposed workers are at an elevated risk of experiencing impaired work performance and cognitive function leading to a greater risk of work-related injuries which includes traumatic injury and a myriad of pathophysiological conditions (e.g., heat stroke, acute kidney injury, adverse cardiovascular events). To mitigate the adverse health effects of occupational heat stress, safety organizations recommend upper limits for heat stress, typically defined by a worker's metabolic rate and the prevailing wet-bulb globe temperature (WBGT). In instances where the heat load created by the combination of work intensity, environment, and clothing worn exceed the upper heat stress limits (uncompensable heat stress), controls such as rest breaks are prescribed to limit increases in core temperature beyond recommended limits. While workers are encouraged to find shelter from the heat during a rest break, it is not always possible or feasible. Typically, workers may rest while remaining exposed to the heat, recover in a shaded area or rest in an air-conditioned room or vehicle. However, the effectiveness of these cooling strategies in mitigating the level of physiological strain experienced by the worker during prolonged work in a hot environment remains unclear. In this project, the investigators will assess the efficacy of the different cooling strategies in preventing excursions in core temperature beyond recommended limits (38.0°C) following the initial stay time for moderate-intensity work in hot ambient conditions (WBGT of 29°C; represents hot outdoor conditions experienced by workers in summers in Ontario, Canada) in context of the prescribed American Conference of Governmental Industrial Hygienists (ACGIH) work-to-rest allocation for unacclimated adults. On three separate days, participants will walk on a treadmill at a fixed metabolic rate of 200 W/m2 until core temperature reaches and/or exceeds 38.0°C or until volitional fatigue. Thereafter, participants will complete an additional 180 min work bout employing the recommended ACGIH work-to-rest allocation of 1:3 (starting with a 45 min rest break followed by a 15 min work bout, with the cycle repeated three times over the 180 min work simulation bout) without (Control) or with cooling mitigation during each 15-min break consisting of either: i) partial cooling equivalent to sitting in a shaded space (WBGT 24°C; 31.7°C and 35% RH) such as under a tree with a light breeze (simulated with pedestal fan fixed at ~2 m/s) or ii) full cooling equivalent to sitting in air-conditioned space (e.g., room or vehicle) maintained at 22°C and 35% RH (equivalent WBGT of 16°C).

ELIGIBILITY:
Inclusion Criteria:

* young (18-30 years) and older adults (50-69 years)
* habitually active, not endurance trained (<2 sessions per week, <150 minutes per week)
* non-smoking
* English or French speaking
* ability to provide informed consent

Exclusion Criteria:

* pre-existing health conditions (e.g., diabetes, hypertension)
* use of medication deemed to significantly modulate thermoregulatory function and heat tolerance (e.g., antidepressants, antihistamines, diuretics)
* engaged in jobs and/or activities that involve frequent exposure to hot environments (e.g., regular sauna use)

Ages: 18 Years to 69 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2024-09-27 (Actual); Primary Completion 2025-03-29 (Actual); Study Completion 2025-03-29 (Actual)

PRIMARY OUTCOMES:
Initial stay time | End of continuous work bout as defined when core temperature reaches 38.0°C or when the maximum of 240 minutes of continuous exercise is achieved
  Total continuous work time to achieve an initial absolute increase in core temperature of 38°C (equivalent to a 1°C increase in body core temperature above resting levels) (note: in instances where a participant voluntarily terminates work prematurely before the absolute core temperature of ≥38°C (or relative increase of ≥1°C) is achieved or the absolute core temperature is <38°C (or relative increase of <1°C), the time of termination or end of the work bout will be taken as the initial stay time respectively).
Average core temperature during work-rest allocations | Period of work-rest allocations over a 180 minute following the initial stay time
  Average core temperature following initial stay time
Heart rate at initial stay time | End of continuous work bout as defined when core temperature reaches 38.0°C or when the maximum of 240 minutes of continuous exercise is achieved
  Heart rate at the initial increase in absolute core temperature of 38°C (or relative increase of 1°C)
Average heart rate during work-rest allocations | Period of work-rest allocations over a 180 minute following the initial stay time
  Average heart rate following initial stay time
Skin temperature at initial stay time | End of continuous work bout as defined when core temperature reaches 38.0°C or when the maximum of 240 minutes of continuous exercise is achieved
  Skin temperature measured at the initial increase in absolute core temperature of 38°C (or relative increase of 1°C)
Average skin temperature during work-rest allocations | Period of work-rest allocations over a 180 minute following the initial stay time
  Average heart rate following initial stay time
Thermal comfort scale at initial stay time | End of continuous work bout as defined when core temperature reaches 38.0°C or when the maximum of 240 minutes of continuous exercise is achieved
  Thermal comfort assessed via a visual analog scale ("How comfortable does your body temperature feel?") (4: very uncomfortable to 1: comfortable)
Thermal comfort scale during work-rest allocations | Period of work-rest allocations over a 180 minute following the initial stay time
  Thermal comfort assessed via a visual analog scale ("How comfortable does your body temperature feel?") (4: very uncomfortable to 1: comfortable)
Thirst sensation scale at initial stay time | End of continuous work bout as defined when core temperature reaches 38.0°C or when the maximum of 240 minutes of continuous exercise is achieved
  Assessed via a visual analog scale ("How thirsty are you?") (9: very, very thirsty to 1: Not thirsty at all)
Thirst sensation scale during work-rest allocations | Period of work-rest allocations over a 180 minute following the initial stay time
  Assessed via a visual analog scale ("How thirsty are you?") (9: very, very thirsty to 1: Not thirsty at all)
Rating of Perceived Exertion at initial stay time | End of continuous work bout as defined when core temperature reaches 38.0°C or when the maximum of 240 minutes of continuous exercise is achieved
  Perceived exertion assessed via a self-report questionnaire upon verbal prompting (6: no exertion at all to 20: maximal exertion).
Rating of Perceived Exertion during work-rest allocations | Period of work-rest allocations over a 180 minute following the initial stay time
  Perceived exertion assessed via a self-report questionnaire upon verbal prompting (6: no exertion at all to 20: maximal exertion).
Orthostatic Intolerance Symptoms Assessment | At the end of the 180 minute work-rest allocations
  Cumulative sum of scores on 6 questions asking participant to rank symptoms associated with orthostatic intolerance. All symptoms scored on a scale from 0 (none) to 10 (worst possible) and include feelings of: (1) "dizziness, lightheadedness, feeling faint, or feeling like you might black out"; (2) "Problems with vision (blurring, seeing spots, tunnel vision, etc.)"; (3) "Weakness"; (4) "Fatigue"; (5) "Trouble concentrating"; and (6) "Head and neck discomfort"

CONTACTS AND LOCATIONS:
Locations (1):
- University of Ottawa, Ottawa, Ontario, Canada